CLINICAL TRIAL: NCT05320289
Title: Feasibility Study of the AblaCare System in Transvaginal Ablation of Ovarian Tissue Under ULTRAsound Visualization in Women With Infertility Due to Polycystic Ovary Syndrome
Acronym: ULTRA-US
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: May Health (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ULTRA-US
Record Dates: First submitted 2022-03-18; First posted 2022-04-11 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Polycystic Ovary Syndrome; Infertility, Female
Keywords: PCOS; Infertility related to PCOS; Ovulation restoration
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- AblaCare Procedure (Experimental): AblaCare Procedure performed with use of the AblaCare Kit intended for transvaginal ablation of ovarian tissue under ultrasound visualization in women with infertility due to polycystic ovary syndrome.
  Interventions: Device: AblaCare System

INTERVENTIONS:
Device: AblaCare System — The intervention includes the short-term use of the AblaCare System, which is comprised of three elements: (1) the AblaCare Needle-Catheter Ablation Device (NCAD) (the Device) a 16G echogenic needle including a bipolar temperature-controlled RF ablation catheter which is clipped and secure onto a vaginal ultrasound probe; (2) the AblaCare Adapter which is clipped onto the ultrasound probe; and (3) the AblaCare Generator: a bipolar radiofrequency (RF) ablation platform utilizing the single use AblaCare NCAD for ovarian tissue ablation.
  Once th patient is under conscious sedation, the physician guides the AblaCare system transvaginally with the use of a transvaginal ultrasound. Once the AblaCare device is safely and securely positioned, the physician will deliver radio frequency energy inside the ovary in order to ablate the tissue.

SUMMARY:
The objective of the study is to provide preliminary evidence for the safety and effectiveness of the AblaCare System in transvaginal ablation of ovarian tissue under ultrasound visualization in women with infertility due to polycystic ovary syndrome (PCOS) who have not responded to first-line ovulation induction treatment or are contraindicated for or decline such treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18 to ≤ 40 years
2. Diagnosis of Polycystic Ovary Syndrome (PCOS) according to Rotterdam criteria: Infertility associated with chronic anovulation or oligomenorrhea, AND EITHER:

   2.1. Ultrasonographic evidence of PCOS (ovarian volume ≥ 10ml and/or ovarian antral follicle count per ovary ≥ 20) OR 2.2. Evidence of hyperandrogenaemia: either clinical (hirsutism defined as mFG level ≥ 4-6 depending on ethnicity) or biochemical (raised serum concentration of androgens (testosterone ≥ 2.5nmol/l, or FAI > 4)
3. At least one ovary with ovarian volume ≥ 10ml
4. Ovarian accessibility: determined by ability to bring transvaginal ultrasound transducer into close proximity to ovaries
5. Failure to respond to first-line pharmacological treatment or is contraindicated for or decline such treatment.
6. At least one patent fallopian tube and normal uterine cavity as determined by sonohysterogram, hysterosalpingogram, or hysteroscopy/laparoscopy within the last 3 years
7. Willing to comply with Clinical Investigation Plan-specified follow-up evaluation
8. Ability to understand study requirements and has sufficient fluency in one of the IRB-approved written translation of the Patient Information and Informed consent form
9. Signed informed consent
10. Normal sperm parameters based on WHO 2010 criteria (concentration ≥ 15 million/mL, total motility ≥ 40%, normal morphology ≥ 4%) within the last year
11. Ability to have regular vaginal intercourse during the study
12. No previous sterilization procedures (vasectomy, tubal ligation) that have been reversed

Exclusion Criteria:

1. Current pregnancy
2. Marked obesity, BMI > 40
3. Marked hyperandrogenism (FAI > 15)
4. Patient is currently participating in another investigational drug or device study that clinically interferes with the endpoints of this study
5. Patient not willing to stop all concomitant first-line oral medications at least 6 weeks prior to study procedure and until the 3-month endpoint is reached, and all other forms of ovulation-induction treatment until the 6-month endpoint is reached
6. Lack of capacity to give informed consent
7. Lack of capacity to follow Clinical Investigation Plan and study requirements including all study follow-up visits
8. Previous ovarian surgery: laparoscopic ovarian drilling, endometriosis surgery, ovarian cysts surgery
9. Patient with known or suspected periovarian adhesions
10. Transvaginal ultrasound transducer cannot be brought into proximity of both ovaries

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
Occurrence of at least one (1) ovulation between treatment and 3-month visit. | 3 months

SECONDARY OUTCOMES:
Occurrence of at least one (1) ovulation between treatment and the 6-month visit with or without 1st line medication 3 months or more post-procedure | 6 months
Successful completion of a complete ovarian tissue ablation procedure, which is defined as achievement of the desired number of ablations within each ovary under ultrasound visualization. | During procedure

OTHER OUTCOMES:
Pain level after procedure completion measured by a Visual Analog Scale (VAS) from 0 (no pain) to 10 (worst pain) | Immediately after procedure completion, at 7-day and at 30-day follow up
Pain medication taken during procedure and after procedure | During procedure, at 7-day and at 30-day follow up
Documented ovulation | Between week 2 and week 24 post-procedure
Documented pregnancy | Between week 2 and week 24 post-procedure, at any point during the study
Menstruation occurrences | From 3-month prior to baseline examination, at 7-day, 30-day, 3-, 6-, 9-, and 12-month follow up
Fertility treatment taken | Up to 12 months
Intercourse activity frequency | At 7- and 30-day, 3-, 6-, 9- and 12-month follow up
Number of ablations performed per ovary and estimated achieved ablation % of total ovary volume | At procedure
Time required to complete procedure, defined as time from first insertion of the ultrasound probe and AblaCare NCAD to the completion of the final ablation | At procedure
Device performance of the AblaCare System, defined as a successful completion of a full ovarian tissue ablation procedure without device deficiency related to one component of the AblaCare system | At procedure
Ovarian volume in mL | At baseline, 3-week, 3-month and 6-month follow up
Ovarian antral follicle count per ovary | At baseline, 3-week, 3-month and 6-month follow up
Ovary morphology: either defined as PCOS or not | At baseline, 3-week, 3-month and 6-month follow up
AMH in pmol/l | At baseline, 3-month and 6-month follow up
Testosterone in nmol/l | At baseline, 3-month and 6-month follow up
Androstenedione in nmol/l | At baseline, 3-month and 6-month follow up
LH in IU/l | At baseline, 3-month and 6-month follow up
FSH in IU/l | At baseline, 3-month and 6-month follow up
Free Androgen Index calculated as the ratio of total Testosterone in nmol/l divided by SHBG in nmol/l and multiplied by 100 | At baseline, 3-month and 6-month follow up
Sex Hormone-Binding Globulin (SHBG) in nmol/l | At baseline, 3-month and 6-month follow up
Menstrual cycle pattern reported as regular, oligomenorrhea or amenorrhea | From 3-month prior to baseline examination, at 7-day, 30-day, 3-, 6-, 9-, and 12-month follow up
Hirsutism evaluation | At baseline, 3-month and 6-month follow up
Acne evaluation | At baseline, 3-month and 6-month follow up
BMI | At baseline, 3-month and 6-month follow up
Quality of life measure by the health-related Quality-of-Life Questionnaire for Women with PCOS at baseline | At baseline, 3-month and 6-month follow up

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oklahoma, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No